CLINICAL TRIAL: NCT00779493
Title: Study Title: Curcumin (Tumeric) in the Treatment of Irritable Bowel Syndrome: A Randomized-Controlled Trial
Brief Title: Curcumin (Tumeric) in the Treatment of Irritable Bowel Syndrome: A Randomized-Controlled Trial
Acronym: CuTIBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4893
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; constipation; diarrhea; gas; bloating; abdominal pain; disturbance of defecation; irritable colon
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Diarrhea; Mucopolysaccharidosis IV; Abdominal Pain | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Curcumin 900mg twice daily by mouth
  Interventions: Dietary Supplement: curcumin
- B (Placebo Comparator): Placebo capsule to be made by Swanson Vitamins to simulate the capsule.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: curcumin — curcumin 900mg twice daily by mouth
  Other Names: Swanson vitamins-curcumin
  Arms: A
Dietary Supplement: placebo — placebo capsule to simulate 900mg curcumin capsule
  Other Names: Swanson curcumin placebo
  Arms: B

SUMMARY:
Evidence exists to support low-grade inflammation as the inciting factor leading to visceral hypersensitivity and alteration in motility in irritable bowel syndrome.In the medical literature,there is ample in vitro and in vivo evidence supporting turmeric and its derivative curcumin as an antitumor, anti-inflammatory and antioxidant agent. We propose a randomized, placebo-controlled, double blinded, parallel treatment study evaluating the effects of turmeric on the symptoms of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

Patients from the hospitals and clinics of the Southern California Permanente Medical Group who conform to the Rome III criteria and

* Age 18 years and above,
* Male or female,
* Able to give consent and follow the treatment plan and be able to answer surveys.
* Negative serum pregnancy test (females of childbearing potential only) and are willing to use an adequate method of contraception throughout the duration of the study.

Exclusion Criteria:

* Any of the following: diabetes, HIV disease, use of anticoagulants or antiplatelet medication, abnormal coagulation or thrombocytopenia, biliary obstruction, inflammatory bowel, symptomatic gallstones, celiac disease, ongoing use of medications known to cause or exacerbate symptoms of IBS and chronic, daily users of IBS medications.
* Use of scheduled IBS medications for 4 weeks prior to and during the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Disease severity will be assessed using the irritable bowel severity score (IBSS) which utilizes a visual analog scale (VAS) (28). The primary outcome will be defined as at least 50% reduction in IBSS. | at 6 months of treatment

SECONDARY OUTCOMES:
Changes in bowel movement frequency, consistency, frequency of as-needed medication use and bloating as measured by the VAS, and improvement SF-36 Quality of Life survey. | end of observation and the end of treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: chris n conteas, md, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States